CLINICAL TRIAL: NCT02834650
Title: Validating Cardiac MRI Biomarkers and Genotype-Phenotype Correlations for Duchenne Muscular Dystrophy (DMD)
Brief Title: Validating Cardiac MRI Biomarkers and Genotype-Phenotype Correlations for DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Children's Hospital of Orange County (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Ennis, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DMD2016; 1R01HL131975-01 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Contrast Media; Hematologic Tests; Heart Rate; Respiratory Physiological Phenomena; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1a (Experimental): Group 1a comprises healthy volunteers who will complete a Cardiac MRI without contrast. A subset of healthy volunteers will have a repeat MRI at Children's Hospital of Orange County.
  Interventions: Other: Cardiac MRI without contrast; Other: Repeat MRI scan
- Group 1b (Experimental): Group 1b comprises boys with DMD who will complete a Cardiac MRI with contrast, a blood test, a heart rate test and a pulmonary function test.
  A subset of boys with DMD will have a repeat MRI with contrast at Children's Hospital of Orange County.
  Interventions: Other: Cardiac MRI with contrast; Other: Blood Test; Other: Heart Rate; Other: Pulmonary Function Test; Other: Genetic Testing; Other: Repeat MRI scan
- Group 2 (Experimental): Group 2 comprises boys with DMD who will complete a Cardiac MRI with contrast, a blood test, a heart rate test and a pulmonary function test and a repeat MRI scan with contrast at 6 Months.
  Interventions: Other: Cardiac MRI with contrast; Other: Blood Test; Other: Heart Rate; Other: Pulmonary Function Test; Other: Genetic Testing; Other: Repeat MRI scan
- Group 3 (Experimental): Group 3 comprises boys with DMD who will complete a Cardiac MRI with contrast, a blood test, a heart rate test and a pulmonary function test and a genetic testing.
  Interventions: Other: Cardiac MRI with contrast; Other: Blood Test; Other: Heart Rate; Other: Pulmonary Function Test; Other: Genetic Testing

INTERVENTIONS:
Other: Cardiac MRI with contrast — Cardiac MRI
  Arms: Group 1b; Group 2; Group 3
Other: Cardiac MRI without contrast — Cardiac MRI
  Arms: Group 1a
Other: Blood Test — Hematocrit, Creatinine, Troponin, BNP
  Arms: Group 1b; Group 2; Group 3
Other: Heart Rate — Holter Monitor
  Arms: Group 1b; Group 2; Group 3
Other: Pulmonary Function Test — Pulmonary Function Test
  Arms: Group 1b; Group 2; Group 3
Other: Genetic Testing — Genetic Testing
  Arms: Group 1b; Group 2; Group 3
Other: Repeat MRI scan — Repeat MRI scan
  Arms: Group 1a; Group 1b; Group 2

SUMMARY:
This study will collect MRI from healthy volunteer boys and boys with Duchenne Muscular Dystrophy (DMD) to help researchers identify and validate cardiac MRI biomarkers to better understand the health of the heart and changes in heart health over time in boys with DMD.

Currently, there is a lack of sufficiently well characterized cardiac MRI biomarkers that can serve as endpoints for detecting on-target and/or off-target cardiac effects during clinical drug trials for boys with DMD.

Consequently, the first objective is to identify and characterize several cardiac MRI biomarkers for boys with DMD.

DETAILED DESCRIPTION:
The second objective is to use their well-characterized cardiac MRI biomarkers and define their sensitivity for detecting early cardiac involvement. The final objective is to use these validated cardiac MRI biomarkers to better understand the genotype-phenotype correlation in boys with DMD, which to date remain tenuous. The investigators propose a pilot study to explore cardiac genotype-phenotype correlations in boys with DMD and outlier phenotypes using approaches they have pioneered for skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy boys or pediatric patients with DMD age 7 to 21
* Able & willing to complete an approximately 75-minute (or less) MRI exam without sedation or mechanical ventilation
* Drug regimen (if applicable) stable for at least 3 months prior to participation

Exclusion Criteria:

* Renal insufficiency (GFR<40 mL/min/m2)
* Non-MRI compatible implants (e.g. neurostimulator, pacemaker, implanted cardioverter defibrillator)
* Claustrophobia that prevents an MRI exam
* Known allergy to MRI contrast agents
* Serum potassium level of >5.0 mmol/L
* Signs and symptoms of heart failure

Ages: 7 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 89 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Myocardial Tissue Characterization | 6 months
  Focal and diffuse fibrosis, intra myocardial fat, edema plus water mobility
Myocardial Functional Characterization | 6 months
  Strain imaging and rotational mechanics
Genomic Analysis | 4 years
  Proposing mechanisms of cardiac dysfunction or protective phenotypes using genomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ennis, PhD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Stanford, California